CLINICAL TRIAL: NCT04610047
Title: A Phase 2b Double-blind, Randomized, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of Norketotifen (NKT) in the Treatment of Acute Uncomplicated Influenza-like Illness (ILI)
Brief Title: Efficacy and Safety of Norketotifen in Uncomplicated Influenza-like Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NKT-203
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Influenza; Influenza -Like Illness
MeSH Terms: conditions — Influenza, Human | interventions — norketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Norketotifen (Experimental): Norketotifen oral capsules, twice daily for 7 days
  Interventions: Drug: Norketotifen
- Placebo (Placebo Comparator): Placebo oral capsules, twice daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norketotifen — Oral capsule
  Arms: Norketotifen
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2b, multi-center, double-blind, randomized, placebo-controlled, parallel-group study of NKT versus placebo in otherwise healthy adults presenting with acute uncomplicated ILI due to influenza or other respiratory viruses in a community setting.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and comply with all study procedures, and willing to provide written informed consent prior to the pre-dose examinations
2. Symptoms of ILI including all of the following:

   * Fever ≥38º Celsius (oral)
   * At least one of the following general systemic symptoms associated with ILI are present with a severity of moderate or greater: headache, feverishness or chills, muscle or joint pain, fatigue
   * At least one of the following respiratory symptoms associated with ILI are present with a severity of moderate or greater: cough, sore throat, nasal congestion
3. Total symptom severity score (sum of the scores of all 7 individual symptoms) of ≥11 in the predose examinations
4. The time interval between the onset of symptoms and the predose examinations is ≤48 hours.
5. Females of childbearing potential and males agree to use an appropriate method of contraception as detailed in the protocol

Exclusion Criteria:

1. Known or suspected infection with Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV2) or Coronavirus Disease 2019 (COVID-19) illness
2. Female subjects who are pregnant, 2 weeks post-partum, or breastfeeding
3. Severe ILI requiring inpatient treatment
4. Any of the following risk factors (according to the CDC's list of People at High Risk for Developing Serious Flu-Related Complications):

   * Extreme obesity (body mass index ≥40 kg/m^2)
   * Residents of nursing homes or other long-term care facilities
   * American Indians and Alaska natives
   * Asthma
   * Chronic lung disease (such as chronic obstructive pulmonary disease or cystic fibrosis)
   * Neurological and neurodevelopmental conditions (including disorders of the brain, spinal cord, peripheral nerve, and muscle such as cerebral palsy, epilepsy [seizure disorders], stroke, intellectual disability, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury)
   * Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease)
   * Blood disorders (such as sickle cell disease)
   * Endocrine disorders (such as diabetes mellitus)
   * Kidney disorders
   * Liver disorders
   * Metabolic disorders (such as inherited metabolic disorders and mitochondrial disorders)
   * Compromised immune system due to disease or medication (such as subjects with human immunodeficiency virus or cancer, or those on chronic steroids)
5. Presence of any severe or uncontrolled medical or psychiatric illness
6. History of or current autoimmune disease
7. History of recurrent lower respiratory tract infection
8. Any concurrent infection requiring systemic antimicrobial and/or antiviral therapy
9. Any clinically significant electrocardiogram (ECG) test
10. Received baloxavir, oseltamivir, peramivir, zanamivir, rimantadine, or amantadine within 30 days prior to the predose examinations
11. Received an investigational monoclonal antibody for a viral disease in the last year prior to the predose examinations
12. Received ketotifen fumarate, cromolyn sodium, or nedocromil sodium by any route of administration within 30 days prior to the predose examinations
13. Exposure to an investigational drug within 30 days prior to the predose examinations
14. History of allergic reaction to ketotifen
15. Any prior exposure to norketotifen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of symptoms | 14 days
  Time to alleviation of the symptoms of ILI (headache, feverishness/chills, muscle/joint pain, fatigue, cough, sore throat, nasal congestion)

SECONDARY OUTCOMES:
Time to resolution of fever (body temperature equal to or less than 37ºC) | 14 days
Proportion of subjects whose symptoms have been alleviated at each time point through Day 14 | 14 days
Change from baseline in composite symptom score at each time point through Day 14 | 14 days
Body temperature at each time point through Day 14 | 14 days
Time to alleviation of individual symptoms (headache, feverishness/chills, muscle/joint pain, fatigue, cough, sore throat, nasal congestion) | 14 days
Time to resumption of normal activity | 14 days
Use of rescue medication (acetaminophen) | 14 days
Time to alleviation of symptoms by confirmed viral pathogen (influenza vs non influenza) | 14 days
Time to resolution of fever by confirmed viral pathogen (influenza vs non influenza) | 14 days

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Precision Trials AZ, Phoenix, Arizona
  - Downtown LA Research Center, Los Angeles, California
  - Omega Research Debary, DeBary, Florida
  - The Chappel Group Research, Kissimmee, Florida
  - South Florida Research Center, Miami, Florida
  - Premier Research Associate, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Horizon Research Group of Opelousas, Eunice, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Relief Integrated Health Care, Louisburg, North Carolina
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Frontier Clinical Research, Scottdale, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Clinovacare Medical Research Center, West Columbia, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinical Research Solutions, Jackson, Tennessee
  - Cedar Health Research, Dallas, Texas
  - Advanced Medical Group, Houston, Texas
  - Frontier Clinical Research, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No